CLINICAL TRIAL: NCT06907030
Title: Evaluation of Operational Wear and Tear Related to the Caledonian Crisis on Military Personnel
Brief Title: Wear and Tear on Military Personnel Post Caledonian Crisis
Acronym: U-CARE
Status: Recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Collaborators: Institut de recherche biomédicale des armées (IRBA), Bretigny sur Orge, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024PPRC08; 2024-A02433-44 (Other: (IDRCB))
Record Dates: First submitted 2025-03-13; First posted 2025-04-02 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Chronic Stress Disorder
Keywords: operational wear and tear; resilience; organisational and human factor; psychosocial risk
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- exposed group: Exposed group is the group of military personnel present in New Caledonia at the start of the crisis, i.e. in May 2024, and still posted to New Caledonia at the time of the study, i.e. in April 2025.
  Interventions: Other: No intervention
- control group: Control group is the group of military personnel not present in New Caledonia at the start of the crisis, i.e. in May 2024, posted to New Caledonia in the summer of 2024 and present at the time of the study, i.e. in April 2025.

INTERVENTIONS:
Other: No intervention — No intervention
  Groups: exposed group

SUMMARY:
Since May 2024, New Caledonia has been experiencing a period of crisis. The organisation of the work of military personnel on the ground has been heavily impacted, with longer working hours, shorter rest periods and increased stress levels (uncertainty about the situation, lack of visibility, etc.).

Prolonged exposure to stress is accompanied by neuronal damage (Ramdani et al., 2024) and operational fatigue, a mindset that results from reversible neuronal damage and appears to be distinct from exhaustion. The aim of this study is to assess the impact of the crisis on the level of operational fatigue. In addition, identifying the organisational and human factors (Jaspers et al., 2024) that may have been protective against operational fatigue could help to optimise the way in which these factors are taken into account in the event of future crises, in order to promote resilience.

DETAILED DESCRIPTION:
Military personnel face specific operational constraints related to their activity. These constraints require physiological adaptation, which can lead to overall biological wear and tear. In our case, the term 'operational wear and tear' refers to the mindset or mental state induced by operational constraints and the chronic stress they impose.

The soldiers deployed in New Caledonia since the riots in May 2024 have had to cope with operational constraints linked to their job, as well as those linked to the insurrection situation. By modifying the physical constraints (longer working hours, less sleep, etc.) and psychological constraints (for example, the unknown duration of the crisis), the current crisis in New Caledonia may have increased operational wear and tear.

The investigators hypothesise that soldiers present in New Caledonia when the riots began have accumulated additional stress related to the crisis and that this could result in greater operational wear and tear than soldiers transferred to New Caledonia in the summer of 2024. However, it is possible that the stress of moving to New Caledonia will counterbalance this effect. For this reason, the study is being conducted over 2 months, in order to assess the evolutionary profile of operational wear and tear.

This is a single-centre observational study of healthy military personnel in New Caledonia. Subjects will be volunteers and their participation or non-participation will not influence their ability to serve, their promotion or their career. Their superiors will not be informed of their participation or non-participation.

Military personnel will be given an oral presentation of the study. On this occasion, the information note will be distributed to them. If they are volunteers, they will have an inclusion visit, notify their non-objection and fill in the first questionnaire. Between two months later, they will complete the second questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* be a member of the military
* be permanently posted to NC at the time of the study

Exclusion Criteria:

* Be on temporary assignment in NC at the time of the study
* Subjects covered by articles L1121-5 to 1121-8 of the Public Health Code, i.e. :

  * Pregnant women, women in labour and nursing mothers
  * Persons deprived of their liberty by judicial or administrative decision
  * Persons subject to psychiatric monitoring under articles L3212-1 and L3213-1 who are not covered by the provisions of article L1121-8
  * Persons of full age who are the subject of a legal protection measure or who are unable to express their consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Serving military personnel aged between 18 and 65 posted to New Caledonia at the time of the study, i.e. between April and July 2025.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Assessing operational wear and tear linked to the crisis | the questionnaire will be completed by the military in April 2025, i.e. 23 months after the start of the crisis for the exposed group
  Difference in the Burn-out Assesment Tool (Schaufeli et al., 2019) questionnaire score between exposed and control groups. This questionnaire consists of 23 items, each scored from 1 to 5. The sum of the scores for each item is then divided by 23 to give a final score of between 1 and 5. Subjects can then be classified as green (score < 2.59), orange (2.59 to 3.02) and red (score >3.02). The questionnaire contains sub-scores for 'exhaustion', 'mental distance', 'cognitive impairment', 'emotional impairment', 'psychological complaints' and 'psychosomatic complaints'.

SECONDARY OUTCOMES:
Assessing the impact of the crisis on Burn-out Assesment Tool sub-scores | Military personnel will complete the questionnaires in April 2025 and June 2025, i.e. there will be a two-month gap between the two sessions.
  Comparison of variations in Burn-out Assesment Tool sub-scores (Schaufeli et al., 2020) between the 'exposed' and 'unexposed' groups and the first and second questionnaire two month later. This questionnaire consists of 23 items, each scored from 1 to 5. The sum of the scores for each item is then divided by 23 to give a final score of between 1 and 5. Subjects can then be classified as green (score < 2.59), orange (2.59 to 3.02) and red (score >3.02). The questionnaire contains sub-scores for 'exhaustion', 'mental distance', 'cognitive impairment', 'emotional impairment', 'psychological complaints' and 'psychosomatic complaints'.
Assessing the benefits of raising awareness of organisational and human factors on operational wear and tear | Military personnel will complete the questionnaires in April 2025 and June 2025, i.e. there will be a two-month gap between the two sessions.
  Comparison of variations of the scores of the Burn-out Assesment Tool between the group sensitised to organisational and human factors and the group not sensitised to organisational and human factor on the first and second questionnaires.
  This questionnaire consists of 23 items, each scored from 1 to 5. The sum of the scores for each item is then divided by 23 to give a final score of between 1 and 5. Subjects can then be classified as green (score < 2.59), orange (2.59 to 3.02) and red (score >3.02). The questionnaire contains sub-scores for 'exhaustion', 'mental distance', 'cognitive impairment', 'emotional impairment', 'psychological complaints' and 'psychosomatic complaints'.
Determining the protective and vulnerability factors (such as Psychosocial Risks) to operational wear and tear | Military personnel will complete the questionnaires in April 2025
  Search for correlations between scores on the Copenhagen Psychosocial Questionnaire (Kristensen et al., 2005) and Burn-out Assesment Tool scores. Burn-out Assesment Tool questionnaire consists of 23 items, each scored from 1 to 5. The sum of the scores for each item is then divided by 23 to give a final score of between 1 and 5. Subjects can then be classified as green (score < 2.59), orange (2.59 to 3.02) and red (score >3.02). The questionnaire contains sub-scores for 'exhaustion', 'mental distance', 'cognitive impairment', 'emotional impairment', 'psychological complaints' and 'psychosomatic complaints'. The Copenhagen Psychosocial Questionnaire consists of 22 items, each scored from 1 to 5. The sum of the scores for each item is then divided by 22 to give a final score of between 1 and 5. 1 is the best outcome, 5 is the worth outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- NOUMEA, Noumea, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaspers GJ, Borsci S, van der Hoeven JG, Kuijer-Siebelink W, Lemson J. Escape room design in training crew resource management in acute care: a scoping review. BMC Med Educ. 2024 Jul 30;24(1):819. doi: 10.1186/s12909-024-05753-z. PMID 39080688
- [Background] Kristensen TS, Hannerz H, Hogh A, Borg V. The Copenhagen Psychosocial Questionnaire--a tool for the assessment and improvement of the psychosocial work environment. Scand J Work Environ Health. 2005 Dec;31(6):438-49. doi: 10.5271/sjweh.948. PMID 16425585
- [Background] Ramdani C, Desruelle AV, Vallee N, Ogier M. Neurofilament-light: Impact of chronic stress on brain. Rev Neurol (Paris). 2024 Dec;180(10):1139-1141. doi: 10.1016/j.neurol.2024.08.001. Epub 2024 Sep 10. No abstract available. PMID 39261122
- [Background] Schaufeli WB, Desart S, De Witte H. Burnout Assessment Tool (BAT)-Development, Validity, and Reliability. Int J Environ Res Public Health. 2020 Dec 18;17(24):9495. doi: 10.3390/ijerph17249495. PMID 33352940
- [Background] Klein O., Marchal C. et Van der Linden N. (2008). L'analyse de médiation en psychologie sociale expérimentale : une introduction non technique. Revue électronique de Psychologie Sociale, n°2, pp. 53-62